CLINICAL TRIAL: NCT07396103
Title: Clinical Study of Intermittent Hypoxia Reduction Using PIMUN: Efficacy Proof-of-Concept
Brief Title: Efficacy of PIMUN by Reducing Intermittent Hypoxia Events
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 210406008-3
Record Dates: First submitted 2024-11-06; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-10

CONDITIONS: Preterm; Apnea of Prematurity; Hypoxemia
MeSH Terms: conditions — Premature Birth; Apnea; Hypoxia

STUDY DESIGN:
Intervention Model Description: experimental, randomized, crossover, not blinded, pilot study
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the origin of each intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIMUN (Active Comparator): 48 hours of dorsal stimulation by PIMUN. Continous cardiorespiratory monitorization- Brain NIRS first 24 hours- 4-5 hours of Polysomnogram at the second day. Blood and urine samples at the finish.
  Interventions: Other: Brain NIRS; Other: Polysomnogram; Other: Reactive oxydative species
- 48 hours without PIMUN (Sham Comparator): 48 hours without PIMUN. Continous cardiorespiratory monitorization- Brain NIRS first 24 hours- 4-5 hours of Polysomnogram at the second day. Blood and urine samples at the finish.
  Interventions: Other: Brain NIRS; Other: Polysomnogram; Other: Reactive oxydative species

INTERVENTIONS:
Other: Brain NIRS — 24 hours of Brain regional oxygen saturation by NIRS
Other: Polysomnogram — 4-5 hours of polysomnogram recording
Other: Reactive oxydative species — Blood and urine samples to detect plasma not albumin bound proteins- neuroprostane and isoflurane

SUMMARY:
The goal of this clinical trial is to learn if the use of PIMUN(medical device) works to reduce the intermittent hypoxemia of 24-34 weeks of birth gestational age babies. . It will also learn about the safety of the use of PIMUN. The main questions it aims to answer are:

Does PIMUN lower the time of oxygen saturation under 90%? What medical problems do participants have using PIMUN? Researchers will compare the use of PIMUN during 48 hours to 48 hours of usual treatments (not using PIMUN).

Participants will:

Use/ or not use of PIMUN for a 48 hours period- randomly assigned. Regional brain oxygenation by near infrared spectroscopy (NIRS) monitoring at the first day of each 48 hours period. 4-6 hours of polysomnography at the second day of each intervention. Plasma and urine stress oxygen metabolites at the end of each 48-hours intervention.

DETAILED DESCRIPTION:
Preterm infants frequently experience intermittent hypoxia (IH) events despite current treatments, leading to potential neurodevelopmental and systemic sequelae. Many of these episodes are related to an ineffective respiratory drive, a central component of apnea of prematurity (AOP). Previous research has shown that dorsal and extremity stimulation can elicit spontaneous respiratory effort in preterm infants. Several clinical studies have demonstrated that mechanized stimulation can reduce the number of apneas and the total time of oxygen saturation below 90%, a key indicator of IH severity.

Building on prior work, the investigators developed and optimized a stimulation protocol that reliably triggers effective breathing. This protocol was incorporated into a novel medical device called PIMUN. PIMUN consists of a soft cotton garment with an integrated inflatable dorsal chamber. The system includes hardware that captures and releases ambient air to generate pulsatile dorsal stimulation according to a proprietary software algorithm. The device operates using electro-mechanical energy and has been designed to ensure safety and comfort during neonatal use.

This pilot, randomized, crossover experimental study aims to evaluate whether pulsatile dorsal kinesthetic stimulation delivered by PIMUN can reduce the total duration of intermittent hypoxia (defined as oxygen saturation <90%) in preterm infants. Secondary analyses include evaluation of deeper desaturation thresholds (<85% and <80%), heart rate parameters, frequency and type of apneas, resuscitation needs, supplemental oxygen requirements, oxidative stress markers, sleep architecture, and regional brain oxygen saturation. Risk monitoring will include assessment of thermoregulation, skin integrity, comfort (NIPS scale), and device performance and safety alarms.

Eligible participants will be preterm infants under 34 weeks of gestation, within the first month of life, and not requiring mechanical ventilation. Each subject will undergo two intervention periods (with and without PIMUN) in randomized order, separated by a washout period. Continuous monitoring using cardiorespiratory and sleep recording systems will allow precise measurement of oxygen saturation, apnea characteristics, heart rate, and sleep stages. Blood and urine samples will be analyzed for oxidative stress markers.

The investigators hypothesize that PIMUN stimulation will decrease total time spent under hypoxic thresholds and reduce the duration and frequency of apneic events without compromising safety, thermoregulation, or sleep quality. This study is expected to generate proof-of-concept data supporting the efficacy and safety of pulsatile dorsal stimulation as an adjunctive approach to managing apnea of prematurity.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants with a gestational age at birth <34 weeks
* Age <30 days at the time of enrollment
* Documented diagnosis of apnea of prematurity (AOP)

Exclusion Criteria:

* Currently receiving mechanical ventilation (MV)
* Presence of major congenital malformations
* Clinically unstable or critically ill at the time of screening
* Active sepsis or undergoing treatment for sepsis
* Intraventricular hemorrhage (IVH) Grade > II
* Receiving sedatives or anticonvulsant medications

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Total Time of Oxygen Saturation <90% | 48-hour data baseline versus 48- hour data with PIMUN
  Total cumulative duration (in minutes) that peripheral oxygen saturation (SpO₂) remains below 90%, measured using cardiorespiratory monitoring and oxygen saturation histogram

SECONDARY OUTCOMES:
Total Time of Oxygen Saturation <85% and <80% | 48-hour data baseline versus 48- hour data with PIMUN
  Cumulative time (in minutes) , derived from continuous cardiorespiratory monitoring and polysomnography (PSG)
Neonatal infant pain scale (NIPS) | 48-hour data baseline versus 48- hour data with PIMUN
  The Neonatal Infant Pain Scale (NIPS) is a validated behavioral assessment tool used to evaluate pain or discomfort in neonates. It is based on six observable indicators of distress:
  Parameter Scoring Criteria Facial Expression 0 = Relaxed muscles 1 = Grimace Cry 0 = No cry 1 = Whimper 2 = Vigorous cry Breathing Patterns 0 = Relaxed 1 = Change in breathing (irregular, labored) Arms 0 = Relaxed/neutral 1 = Flexed/extended Legs 0 = Relaxed/neutral1 = Flexed/extended State of Arousal 0 = Sleeping/quiet 1 = Fussy/awake
  Total Score Range: 0-7 0-2: No pain or mild discomfort 3-4: Moderate pain
  ≥5: Severe pain
  Scores are typically assessed by trained nursing staff during clinical or research interventions. The NIPS provides an objective measure of neonatal comfort and can be used to monitor procedural pain, device tolerance, or overall well-being during treatment.
Total Time of Heart Rate <100 bpm | 48-hour data baseline versus 48- hour data with PIMUN
  Total Time of Heart Rate <100 bpm/Cumulative time (in minutes) , measured via continuous ECG monitoring and PSG event extraction
Number of Apnea Events (Central, Mixed, or Obstructive) | 48-hour data baseline versus 48- hour data with PIMUN
  Description: Total count of central, mixed, and obstructive apneas per hour of recording, detected by cardiorespiratory monitoring and PSG.
  Unit of Measure: Events per hour
Duration of Desaturation Episodes | 48-hour data baseline versus 48- hour data with PIMUN
  Length of individual desaturation episodes categorized as <10 seconds, 10-20 seconds, or >20 seconds, obtained from event data extraction.
  Unit of Measure: Seconds per episode
REM and Non-REM Sleep Duration | baseline versus during the use of PIMUN
  Total time spent in REM and non-REM sleep stages, determined from polysomnography recordings.
  Unit of Measure: Minutes
Need for Resuscitation or Respiratory Support | 48-hour data baseline versus 48- hour data with PIMUN
  Frequency of episodes requiring resuscitation, supplemental oxygen, or connection to mechanical ventilation as recorded by nursing staff.
  Unit of Measure: Number of events
Oxidative Stress Marker Levels | baseline versus after 48- hour using PIMUN
  Change in oxidative stress biomarkers (e.g., plasma carbonyls, urinary isoprostanes) from baseline to end of intervention period.
  Unit of Measure: Concentration (e.g., μmol/L or ng/mL)

OTHER OUTCOMES:
Number and type of Safety Events | During each 48-hour intervention period
  Report of any adverse event, defined as any skin reaction- apneas requiring resuscitation- increasing therapy of AOP- connection to MV- thermoregulation disturbances- Device failure- etc.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Clinica San Carlos de Apoquindo, Santiago, Santiago Metropolitan
  - UC Christus Clinical Hospital, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No